CLINICAL TRIAL: NCT00753506
Title: Double-Blind Trial of Artemisinin to Reduce The Symptoms of Schizophrenia
Brief Title: Artemisinin to Reduce The Symptoms of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheppard Pratt Health System (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Faith Dickerson, PhD, MPH, Head, Stanley Research Program, Sheppard Pratt Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMRI/SPHS: 2007-02
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Results first posted 2012-02-20 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — artemisinin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Artemisinin (Active Comparator): 100 mg artemisinin capsule
  Interventions: Dietary Supplement: Artemisinin
- Placebo (Placebo Comparator): Identical looking placebo capsule
  Interventions: Dietary Supplement: Identical looking placebo capsule

INTERVENTIONS:
Dietary Supplement: Artemisinin — 100 mg of artemisinin twice per day for 10 weeks
  Arms: Artemisinin
Dietary Supplement: Identical looking placebo capsule — Identical looking placebo twice per day for 10 weeks
  Arms: Placebo

SUMMARY:
The investigators intend to explore the hypothesis that symptoms of schizophrenia may be reduced by the antimalarial compound artemisinin when used in addition to standard antipsychotic medications.

DETAILED DESCRIPTION:
The aims of the current study are:

1. To evaluate the efficacy and side effects of artemisinin as an add-on compound for patients with schizophrenia who have residual psychotic symptoms of at least moderate severity.
2. To evaluate the effect of artemisinin on cognitive impairments and associated functional skills.
3. To investigate whether treatment with artemisinin produces a significant effect on the levels of antibodies to Toxoplasma.
4. To examine whether changes in cognitive impairment or psychiatric symptoms are correlated with changes in antibodies to Toxoplasma before and during the treatment with artemisinin.

ELIGIBILITY:
Inclusion Criteria

* Age 18-65 years old.
* Capacity for written informed consent.
* Primary Axis I diagnosis (DSM-IV) of schizophrenia, any type, OR schizoaffective disorder (APA, 1994).
* Currently an outpatient at the time of enrollment.
* Residual psychotic symptoms which are at least moderately severe as evidenced by one or more Positive and Negative Syndrome Scale (PANSS) positive symptom scores, and/or PANSS negative symptom scores of 4 or more; OR a total PANSS score of 50 or more, containing at least three positive or negative items with scores of 3 or more at screening.
* Conformance to Patient Outcome Research Team (PORT) Treatment Recommendation #5, Maintenance Antipsychotic Medication Dose (Lehman et al., 2004).
* Receiving antipsychotic medication for at least 8 weeks prior to starting the study with no medication changes within the previous 21 days.
* Participants must be proficient in English.

Exclusion Criteria

* Diagnosis of mental retardation.
* History of IV drug use.
* Any serious medical condition that affects brain or cognitive functioning (e.g., epilepsy, serious head injury, brain tumor or other neurological disorder).
* HIV infection or other immunodeficiency condition.
* Primary diagnosis of substance abuse or dependence according to DSM-IV criteria within the last three months.
* Participated in any investigational drug trial in the past 30 days.
* Pregnancy or planning to become pregnant during the study period.
* Any clinically significant or unstable medical disorder as determined by the investigators that would preclude study participation, including congestive heart failure, abnormal liver function or disease, renal failure, and any diagnosis of cancer undergoing active treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faith B Dickerson, PhD, MPH, Principal Investigator — Stanley Research Program at Sheppard Pratt
Locations (1):
- Sheppard Pratt Health System, Towson, Maryland, United States

REFERENCES:
- [Result] Dickerson F, Stallings C, Vaughan C, Origoni A, Goga J, Khushalani S, Yolken R. Artemisinin reduces the level of antibodies to gliadin in schizophrenia. Schizophr Res. 2011 Jul;129(2-3):196-200. doi: 10.1016/j.schres.2011.04.010. Epub 2011 May 5. PMID 21546216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled n=66 participants drawn from the Sheppard Pratt Health System and from rehabilitation and treatment programs in Central Maryland. Dates of recruitment 8/08-1/10.
Pre-assignment Details: We used a two week placebo run in for all participants
Groups:
- Artemisinin: Artemisinin 100 mg capsule Artemisinin (qinghaosu) is the antimalarial principle isolated by Chinese scientists from Artemisia annua L. (Sweet Wormwood plant), which has been in use in China for more than 2,000 years as an herbal tea against fever (van Agtmael et al., 1999). Artemisinin is a sesquiterpene trioxane lactone with a peroxide bridge linkage and is poorly soluble in oils or water. Johns Hopkins collaborators recently synthesized novel, nonacetal, hydrolytically stable derivatives of artemisinin and showed that they inhibit the replication of Toxoplasma gondii in cell culture (Jones-Brando et al., 2006).
- Placebo: Identical looking placebo capsule The placebo will contain an inert powder which is typically used to make many pharmaceutical tablets. The control capsules will be identical looking to the artemisinin capsules and will be prepared for use in this study by the Temple University Pharmacy which has experience in preparing materials for clinical trials.
Period: Overall Study
Arm/Group | Artemisinin | Placebo
Started | 33 | 33
Completed | 26 | 31
Not Completed | 7 | 2
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other reason | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Artemisinin | Placebo | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 33 | 66
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.4 (9.0) | 49.2 (9.2) | 47.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 20 | 18 | 38
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Score From the Beginning to the End of the Double-blind Treatment Phase Weeks 2-12
Description: The Positive and Negative Syndrome Scale (PANSS) measures psychiatric symptomatology, especially related to psychosis. The complete PANSS contains ratings for 30 symptoms, including 7 positive symptoms, 7 negative symptoms, and 16 general psychiatric symptoms. The severity of each symptom is rated on a scale ranging from 1 (minimal) to 7 (extreme); higher scores indicate increased symptomatology. Total PANSS scores include scores from all categories and range from 30 to 210 units on a scale. PANSS positive symptom scores and negative symptom scores each range from 7 to 49 units on a scale.
Time Frame: 10 weeks (weeks 2 & 12)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Artemisinin: 100 mg capsule of artemisinin taken twice per day.
- Placebo: 100 mg artemisinin identical placebo capsule taken twice per day.
Arm/Group | Artemisinin | Placebo
Number analyzed (Participants) | 26 | 31
units on a scale
  Week 2 PANSS total symptom score | 64 (8.74) | 68.13 (9.07)
  Week 12 PANSS total symptom score | 61.42 (10.53) | 66.32 (9.45)
  Week 2 PANSS positive score | 15.42 (4.18) | 16.26 (3.96)
  Week 12 PANSS positive score | 14.92 (5.11) | 16.35 (5.35)
  Week 2 PANSS negative score | 19.08 (3.12) | 19.77 (3.48)
  Week 12 PANSS negative score | 18.69 (3.69) | 19.03 (3.67)
  Week 2 PANSS general score | 29.5 (5.32) | 32.10 (6.18)
  Week 12 PANSS general score | 27.81 (4.78) | 30.94 (4.84)
Statistical Analysis 1: Comparison: Artemisinin vs Placebo; Repeated measures analaysis of variance; Test type: Superiority or Other; p > 0.10, ANOVA; F = 1.59

2. Secondary Outcome: Change in Cognitive Functioning as Measured by the Repeatable Battery for the Assessment of Neuropsychological Status and Change in Functional Performance as Measured by the UCSD Performance-based Skills Assessment.
Time Frame: 10 weeks (weeks 2 & 12)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8/08-1/10
Arm/Group | Artemisinin | Placebo
Serious Adverse Events (participants affected / at risk) | 3/33 | 3/33
Other Adverse Events (participants affected / at risk) | 0/26 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artemisinin (N=33) | Placebo (N=33)
Arm fracture requiring hospitalization (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Atypical chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Schizophrenia exacerbation (Psychiatric disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No